CLINICAL TRIAL: NCT03941314
Title: A Prospective Randomized, Parallel-group, Multicentre, Superiority Trial of the SUPERA Peripheral Stent System in Patients With Femoro-popliteal Artery Disease
Brief Title: A Superiority Trial of the SUPERA Peripheral Stent System in Patients With Femoro-popliteal Artery Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Abbott (Industry); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2019-00312; CTU 17/037 (Other: CTU Kantonsspital St. Gallen)
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supera® Peripheral Stent System (Experimental): Femoro-popliteal arterial stenting with Supera® Peripheral Stent System as CE-marked by the manufacturer Abbott
  Interventions: Device: Supera® Peripheral Stent System
- EverFlex™ Self-Expanding Peripheral Stent System (Active Comparator): Femoro-popliteal arterial stenting with EverFlex™ Self-Expanding Peripheral Stent System with Entrust™ Delivery System or as Protégé™ EverFlex™
  Interventions: Device: EverFlex™ Self-Expanding Peripheral Stent System

INTERVENTIONS:
Device: Supera® Peripheral Stent System — The index procedure is placing a selfexpandable stent at a femoro-popliteal location. The way the stenosis or occlusion is traversed is not part of the study. It is mandatory to prepare then the vessel with PTA (at least the size of the stent) and thereafter insert the stent. Post-PTA can be performed with same balloon, but post-PTA is not mandatory to be performed.
  Arms: Supera® Peripheral Stent System
Device: EverFlex™ Self-Expanding Peripheral Stent System — The index procedure is placing a selfexpandable stent at a femoro-popliteal location. The way the stenosis or occlusion is traversed is not part of the study. It is mandatory to prepare then the vessel with PTA (at least the size of the stent) and thereafter insert the stent. Post-PTA can be performed with same balloon, but post-PTA is not mandatory to be performed.
  Other Names: EverFlex™ with Entrust™ Delivery System or Protégé™ EverFlex™
  Arms: EverFlex™ Self-Expanding Peripheral Stent System

SUMMARY:
The purpose of this study (superiority trial) is to compare the Supera® Peripheral Stent System with a standard nitinol self-expanding stent for treatment of femoro-popliteal arterial occlusive disease.

Hypothesis:

The Supera® stent is superior to a standard nitinol self-expanding stent, for treatment of femoro-popliteal artery disease in terms of (1) primary patency rate and (2) need for revascularization up to 24 months after stent insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with femoro-popliteal artery disease, who will require a stent femoro-popliteal following failed percutaneous transluminal angioplasty (PTA)
* Target Lesion length <200mm
* Planned follow-up available for at least 24 months
* Written informed consent to participate in the study and agreement to comply with the study protocol must be obtained from the patient prior to initiation of any study-mandated procedure and randomization

Exclusion Criteria:

* Life expectancy <24 months
* Patients who cannot receive dual antiplatelet therapy (aspirin 100mg and clopidogrel 75mg) or anticoagulation therapy
* Patients with known allergies to: nitinol (nickel titanium); or contrast agent, that cannot be medically managed
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Prior stenting at the location of intended stenting
* Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the stent or stent delivery system
* Enrolment of study investigator, his/her family members, employees and other dependent persons
* If female and of childbearing potential: known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Difference in primary patency rate (proportion of patients classed as treatment succsess) | 24 months
  Peak systolic velocity ratio assessed with Duplex ultrasound (Treatment success is defined as Peak Systolic Velocity (PSV) ratio < 2.5 at the stented target lesion measured by Duplex ultrasound (DUS) indicating freedom from >50% restenosis with no clinically driven re-intervention within the stented segment.)

SECONDARY OUTCOMES:
Difference in primary patency rate | 1 month, 6 months, 12 months
  Peak systolic velocity ratio assessed with Duplex ultrasound
Difference in target lesion/vessel revascularization | 24 months
  Patients with target lesion revascularization due to restenosis or target vessel revascularization.
Difference in amputation | 24 months
  Proportion of patients with amputation (minor or major)
Difference in time to restenosis (and time to target lesion revascularization due to restenosis) | 24 months
Difference in Anklre Brachial Index | 1 month, 6 months, 12 months, 24 months
  Ankle Brachial Index of the treated lesion
Difference in Fontaine classification | 1 month, 6 months, 12 months, 24 months
  Fontaine classification

OTHER OUTCOMES:
Rate of site complications [Safety Endpoint] | 1 month
Rate of prolonged hospital stay [Safety Endpoint] | 1 month
Rate of need for surgical revision [Safety Endpoint] | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Binkert, MD, Principal Investigator — Kantonsspital Winterthur KSW
Locations (3):
- Hospital Carlos Haya, Málaga, Spain
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur